CLINICAL TRIAL: NCT00420225
Title: Low-Weight Polypropylene Mesh for Anterior Vaginal Wall Prolapse: A Prospective Randomized Study
Brief Title: Mesh Repair of Anterior Vaginal Wall Prolapse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tampere University Hospital
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Anterior Vaginal Wall Prolapse
Keywords: Cystocele; surgery; mesh; genital prolapse
MeSH Terms: conditions — Cystocele

INTERVENTIONS:
Device: Low-weight prolypropylene mesh

SUMMARY:
The purpose of this study is to determine whether reenforcement with polypropylen mesh compared with traditional anterior colporrhaphy for anterior vaginal wall prolapse results in fewer recurrences.

DETAILED DESCRIPTION:
Anterior vaginal wall prolapse is the most common type of pelvic organ prolapse in postmenopausal women. This anatomic defect has traditionally been repaired with anterior colporrhaphy plication, a series of interrupted stitches being the main surgical component. The procedure is associated with a high recurrence rate, up to 32 % even after using paravaginal repair along with anterior colporrhaphy.It has been sought to resolve the problem of recurrence using artificial mesh as in the repair of abdominal hernias.

Comparison: Anterior vaginal wall repair with or without reinforcement with polypropylene mesh were compared in a prospective randomized study

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with symptomatic anterior vaginal wall prolapse to the hymen or beyond when under strain and referred for reconstructive pelvic surgery

Exclusion Criteria:

* an apical defect indicating concomitant vaginal fixation, or stress urinary incontinence necessitating surgery, or her main symptomatic prolapse component was in the posterior vaginal wall.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202
Dates: Start 2003-04; Study Completion 2008-05

PRIMARY OUTCOMES:
Recurrence of anterior vaginal wall prolapse

SECONDARY OUTCOMES:
Postvoidal residual urine
Symptom resolution
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nieminen, Principal Investigator — Tampere University Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Tampere University Hospital, Department of Obstetrics and Gynaecology, Tampere, Finland

REFERENCES:
- [Derived] Nieminen K, Hiltunen R, Heiskanen E, Takala T, Niemi K, Merikari M, Heinonen PK. Symptom resolution and sexual function after anterior vaginal wall repair with or without polypropylene mesh. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Dec;19(12):1611-6. doi: 10.1007/s00192-008-0707-7. Epub 2008 Aug 21. PMID 18716704